CLINICAL TRIAL: NCT06119243
Title: Multicenter Study of Near Vision Behavior and Outdoor Time in Children Undergoing Myopia Control
Brief Title: Multicenter Evaluation of Near Vision and Outdoor Time in Kids Study
Acronym: MENOK
Status: Recruiting | Type: Observational
Sponsor: The University of New South Wales (Other)
Collaborators: Queensland University of Technology (Other); New England College of Optometry (Other); State University of New York College of Optometry (Other); University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Pauline Kang, Senior Lecturer, The University of New South Wales
Other Study IDs: MENOK
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myopia
Keywords: Myopia; Myopia control; Progressive myopia; Near vision behavior; Outdoor activity; Environment; Light exposure
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Device: Vivior — The Vivior is a wearable clip-on sensor that objectively quantifies near viewing distance and duration, and ambient illumination. The Vivior will be attached to the spectacles frame of children undergoing myopia control treatment.

SUMMARY:
Currently, optical and pharmacological interventions have been developed to prevent the progression of childhood myopia. However, no myopia control strategy has been shown to have complete efficacy in controlling myopia progression in children. One possible reason is that risk factors contributing to the development of myopia were not controlled in previous clinical studies including time outdoors and near vision behaviour. This study aims to quantify time spent outdoors and near vision behavior in myopic children and its impact on myopia control efficacy. The outcomes of this study will guide clinicians on risk management and improve responses to existing treatments for progressive myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 to below 14 years old
2. Spherical equivalent myopic refractive error greater than -0.50 D
3. Best corrected logMAR visual acuity of 0.1 or better in each eye for 6- to 14-year-old children, and 0.2 logMAR or better than in each eye for 4 and 5-year-old children (adjusted for age-related expectations)
4. Good ocular and general health that would not preclude them from myopia control
5. Competent enough in English to fully understand the participant information and consent form
6. Willing to undergo treatment to slow myopia progression for one year

Exclusion Criteria:

1. Strabismus at distance or near, or amblyopia
2. Systemic or ocular conditions that may affect contact lens use (e.g. severe allergy) or refractive development (e.g. ptosis)
3. Previous history of ocular surgery, trauma or chronic ocular disease that may affect their vision
4. Ocular or systemic medication use which may interfere or interact with myopia treatment or ocular development
5. Child, parents or guardians not willing to comply with treatment and/or follow-up schedule and planning to migrate or move during the one-year study duration

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Myopic children will be recruited from the university based myopia control clinic. Some clinical sites have collaborated with community optometry practices so support recruitment.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Near viewing duration | 12 months
  Duration during near tasks
Near viewing distance | 12 months
  Distance during near tasks
Outdoor time | 12 months
  Ambient illumination to determine time spent outdoors

SECONDARY OUTCOMES:
Objective cycloplegic central refraction | 12 months
  Change in objective refraction to measure myopia progression
Axial length | 12 months
  Change in axial length to measure myopia progression
Subjective cycloplegic central refraction | 12 months
  Change in subjective refraction to measure myopia progression

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - School of Optometry, University of California, Berkeley, Berkeley, California
  - New England College of Optometry, Boston, Massachusetts
  - State University of New York (SUNY), College of Optometry, New York, New York
- Australia (2):
  - School of Optometry and Vision Science, UNSW, Sydney, New South Wales
  - Optometry and Vision Science, Queensland University of Technology, Kelvin Grove, Queensland

IPD SHARING:
Plan to Share IPD: No